CLINICAL TRIAL: NCT00002281
Title: An Open Label Phase I/II Study of Recombinant Granulocyte Colony-Stimulating Factor (r-metHuG-CSF) and Recombinant Erythropoietin (rHuEPO) Given Subcutaneously Along With Zidovudine (AZT) to Patients With AIDS or ARC
Brief Title: A Study of Granulocyte Colony-Stimulating Factor Plus Recombinant Erythropoietin Plus Zidovudine in Patients With AIDS or AIDS-Related Complex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amgen (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 061A; GCSF-8808-109
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-01

CONDITIONS: HIV Infections; Cytopenias
Keywords: Injections, Subcutaneous; Erythropoietin; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Cytopenia; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Filgrastim; Epoetin Alfa; Zidovudine

INTERVENTIONS:
Drug: Filgrastim
Drug: Epoetin alfa
Drug: Zidovudine

SUMMARY:
To evaluate the safety, tolerance and biological activity of filgrastim (granulocyte colony-stimulating factor; G-CSF) given by daily subcutaneous (SC) injection prior to and concomitantly with erythropoietin (EPO) and zidovudine (AZT) in patients with AIDS or severe AIDS related complex (ARC). To evaluate the safety, tolerance, and biological activity of EPO given 3 times weekly by SC injection concomitantly with G-CSF and prior to and concomitantly with AZT in patients with AIDS or severe ARC. To study the safety and tolerance of 3 dose levels of AZT given to patients with AIDS or severe ARC concomitantly treated with G-CSF and EPO. To study the effect of G-CSF alone and in combination with EPO on HIV replication in vivo as measured by circulating HIV p24 antigen, plasma HIV viremia and semiquantitative HIV cocultures.

ELIGIBILITY:
Inclusion Criteria

Concurrent Treatment:

Allowed:

* Radiation or laser therapy to Kaposi's sarcoma lesions provided the dose does not exceed 3000 rads to any one lesion group and/or greater than 10 cm2 total body surface area.

Patients must have:

* A diagnosis of AIDS or AIDS related complex (ARC) as defined by current CDC guidelines.
* Life expectancy > 6 months.
* Defined blood cell counts that may be achieved by transfusion.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* History of malignancy other than Kaposi's sarcoma (KS).
* Presence of > 50 cutaneous KS lesions or progression of KS over the previous 30 days.
* Presence of opportunistic infection requiring ongoing therapy with known bone marrow suppressive agents.
* History of cardiovascular disease.
* History of seizures.
* HIV related dementia or altered mental status that would prohibit the giving and understanding of informed consent.
* Presence of iron deficiency anemia as defined by serum ferritin < 30 ng or iron to TIBC ratio < 15 percent.
* A PT > 15 and a PTT > 40 unless due to a documented circulating lupus anticoagulant.

Concurrent Medication:

Excluded:

* Trimethoprim / sulfamethoxazole.
* Fansidar.
* Non-FDA approved antiretrovirals.
* Hyperimmunization with polio virus.
* Ribavirin.
* Isoprinosine.
* Dextran sulfate.
* Fu zheng herbs.
* AL 721 or its congeners.
* Imuthiol.
* Interferons.
* Chronic use of acyclovir (> 10 days out of 30 days).
* = or > 3g/day oral vitamin C.

Patients with the following are excluded:

* Co-existing conditions and symptoms described in Patient Exclusion Co-existing Conditions.

Prior Medication:

Excluded within 2 weeks of study entry:

* Any non-FDA approved drug.
* Excluded within 4 weeks of study entry:
* Systemic cytotoxic chemotherapy for Kaposi's sarcoma.
* Investigational agents.
* Excluded:
* Colony stimulating factors.

Prior Treatment:

Excluded within 4 weeks of study entry:

* Radiation therapy for Kaposi's sarcoma exceeding 3000 rads to any one lesion group and/or greater than 10 cm2 total body surface area.

Risk Behavior:

Excluded within 3 months of study entry:

* Regular excessive use of alcohol, hallucinogens or other psychotropic agents which are possibly addicting.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Med Ctr, Los Angeles, California, United States

REFERENCES:
- [Background] Miles SA, Mitsuyasu RT, Moreno J, Baldwin G, Alton NK, Souza L, Glaspy JA. Combined therapy with recombinant granulocyte colony-stimulating factor and erythropoietin decreases hematologic toxicity from zidovudine. Blood. 1991 May 15;77(10):2109-17. PMID 1709368